CLINICAL TRIAL: NCT04284514
Title: Phase 1 Multi Center, Double-Masked, Randomized, Placebo-Controlled, Multiple Ascending Dose Cohort Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single or Twice Daily Doses of AKB-9778 Ophthalmic Solution
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AKB-9778 Ophthalmic Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aerpio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AKB-9778-CI-OS-1001
Record Dates: First submitted 2019-08-09; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Ocular Hypertension; Primary Open Angle Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AKB-9778 Ophthalmic Solution (Experimental): Up to 4 daily dose levels of AKB-9778 Ophthalmic Solution will be evaluated. Doses will be administered in both eyes daily for 7 days.
  Interventions: Drug: AKB-9778 Ophthalmic Solution
- Vehicle Control Ophthalmic Solution (Placebo Comparator): Matched vehicle-control ophthalmic solution will be administered in both eyes daily for 7 days.
  Interventions: Drug: Placebo Ophthalmic Solution

INTERVENTIONS:
Drug: AKB-9778 Ophthalmic Solution — AKB-9778 Ophthalmic Solution
  Arms: AKB-9778 Ophthalmic Solution
Drug: Placebo Ophthalmic Solution — Matched vehicle-control
  Arms: Vehicle Control Ophthalmic Solution

SUMMARY:
The purpose of this Phase 1b study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of AKB-9778 ophthalmic solution (eye drops) administered for 7 days in adults. The study is a double-masked, multiple- ascending dose trial and will enroll four cohorts of up to 12 subjects. Dose cohorts will receive increasing doses of AKB-9778 ophthalmic solution or vehicle-matched placebo daily for 7 days. Cohort 5 will enroll subjects with open angle glaucoma or ocular hypertension who will continue current prostaglandin therapy during the study. Cohort 5 subjects will receive the maximum tolerated dose from the previous cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

* Aged > 18 years to 70 years inclusive in Cohort 1; aged ≥ 45 to 70 years inclusive in Cohorts 2-4, aged 18 to 80 years inclusive in Cohort 5.
* For subjects in Cohort 1, IOP between 12 and 23 mm Hg (inclusive). For subjects in Cohorts 2-4, IOP between 16 and 23mm Hg (inclusive). For subjects in Cohort 5, IOP between 17 and 27 mm Hg (inclusive).
* Central corneal thickness of 480 to 600 μm, inclusive
* For subjects in Cohort 5, diagnosis of OAG or OHT
* For subjects in Cohort 5, currently receiving prostaglandin therapy for IOP lowering

Key Exclusion Criteria:

* Diagnosis of any form of glaucoma in Cohorts 1-4
* Clinically significant eye trauma within 6 months of screening
* Any intraocular ophthalmic procedure within 6 months of screening
* Any ocular inflammation within 90 days of screening or a history of recurrent uveitis in either eye
* Subjects with any known chronic ocular disease (other than incipient cataract or refractive error)
* Any condition preventing valid applanation tonometry measurement, e.g., clinically significant corneal disease, refractive surgery
* Visual acuity (VA) worse than 20/30 in either eye, For Cohort 5 VA worse than 20/100 in either eye

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Baseline to Day 7
Vital sign- systolic and diastolic blood pressure | Baseline to Day 7
  Systolic and diastolic blood pressure in mmHg
Complete blood count | Baseline to Day 7
  White blood cells with differential, hemoglobin, hematocrit and platelet count

SECONDARY OUTCOMES:
Intraocular pressure | Baseline to Day 7
  Intraocular pressure in mmHg
AKB-9778 concentration | Baseline to Day 7
  Measurement of AKB-9778 in plasma after drug administration

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - PPD, Austin, Texas
  - Covance Clinical Research Unit, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No